CLINICAL TRIAL: NCT02536768
Title: Evaluation of the National Department of Health's National Adherence Guidelines for Chronic Diseases in South Africa Using Routinely Collected Data
Brief Title: Evaluation of South Africa's National Adherence Strategy
Acronym: ENHANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: World Bank (Lead institution) (Unknown); Republic of South Africa National Department of Health (Lead institution) (Unknown)
Responsible Party: Principal Investigator, Matthew Fox, Professor (Note: Not the PI, but one Co-PI), Boston University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-34074; 7173709 (Other Grant/Funding Number: World Bank)
Record Dates: First submitted 2015-08-26; First posted 2015-09-01 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: HIV; Tuberculosis; Diabetes; Hypertension
Keywords: Medication adherence; ART; Counseling; Adherence Guidelines for Chronic Diseases (HIV, TB and NCDs)
MeSH Terms: conditions — Tuberculosis; Diabetes Mellitus; Hypertension; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Minimum package of interventions to improve ART adherence including fast track initiation counselling, decentralized drug delivery, adherence clubs, fast patient tracing and spaced visits
  Interventions: Behavioral: Minimum package of interventions to improve ART adherence
- Comparison (No Intervention): Standard of care HIV treatment

INTERVENTIONS:
Behavioral: Minimum package of interventions to improve ART adherence — Package of 5 interventions to antiretroviral therapy adherence including fast track initiation counselling, decentralized drug delivery, adherence clubs, fast patient tracing and spaced visits
  Arms: Intervention

SUMMARY:
NOTE THAT THE STUDY IS LED BY SOUTH AFRICA NATIONAL DEPARTMENT OF HEALTH AND WORLD BANK WITH SUPPORT FROM BOSTON UNIVERSITY. The South Africa National Department of Health (NDOH) intends to launch its newly developed National Adherence Guidelines for Chronic Diseases (HIV, TB and NCDs) throughout South Africa in the coming year. Early implementation of the "minimum package" of interventions described in the Adherence Guidelines for HIV patients will take place at 12 primary health clinics and community health centres in four provinces starting in July 2015. To maximize the learning potential of this early implementation stage, NDOH will match the intervention clinics with 12 comparison clinics and randomly allocate intervention or comparison status within the pairs of clinics. This will allow the outcomes of the interventions to be evaluated using a cluster-randomized design and generate data on the costs of implementation and the potential need for adherence support for the other diseases addressed in the guidelines (tuberculosis, hypertension, and diabetes). This protocol is for the evaluation, which will generate information on the effectiveness of minimum package interventions and help improve the design, implementation, and budgeting of the guidelines.

DETAILED DESCRIPTION:
The study will assess the effectiveness of five interventions in the minimum package: 1) Fast track initiation counseling for patients eligible for antiretroviral therapy; 2) Enhanced adherence counseling for unstable patients on HIV treatment; 3) adherence clubs for stable patients on HIV treatment; 4) decentralized medication delivery for stable patients on HIV treatment; and 5) early tracing of all patients who miss an appointment by two weeks. This study will also estimate for each study site an overall "adherence guideline impact" to provide an indication of the effectiveness of the package as a whole.

In addition, the study will estimate the cost of each of the interventions listed above compared to standard of care. Finally, the study will describe the cascade of care for tuberculosis, hypertension, and diabetes, three other chronic diseases for which little information currently exists. To evaluate these interventions the study team will work with the National Department of Health (which will implement the interventions) to randomize 24 clinics in 4 provinces 1:1 to receive the interventions or continue standard of care. All evaluations will use data routinely collected by the clinics, with no study interaction with subjects. A total of 8,256 patients will be enrolled and followed for up to 20 months to estimate short- and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Meet the inclusion criteria for one or more intervention
* Not resident in the facility's catchment area
* Recorded intention to transfer care to a different facility within 12 months

Exclusion Criteria:

* Pregnant and eligible for PMTCT

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8020 (Actual)
Dates: Start 2015-09; Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Alive and in care using clinical records | 3-12 months
  Patient has attended the clinic between 3 and 12 months after being eligible for an intervention
HIV viral supression using lab data | 4-12 months
  HIV viral load measure below 400 copies per ml between 4 and 12 months after eligibility for an intervention

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Fox, DSc, Principal Investigator — Boston University
Locations (1):
- Johannesburg Site, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Larson BA, Pascoe SJS, Huber A, Long LC, Murphy J, Miot J, Fraser-Hurt N, Fox MP, Rosen S. Fast-track treatment initiation counselling in South Africa: A cost-outcomes analysis. PLoS One. 2021 Mar 18;16(3):e0248551. doi: 10.1371/journal.pone.0248551. eCollection 2021. PMID 33735206
- [Derived] Pascoe SJS, Scott NA, Fong RM, Murphy J, Huber AN, Moolla A, Phokojoe M, Gorgens M, Rosen S, Wilson D, Pillay Y, Fox MP, Fraser-Hurt N. "Patients are not the same, so we cannot treat them the same" - A qualitative content analysis of provider, patient and implementer perspectives on differentiated service delivery models for HIV treatment in South Africa. J Int AIDS Soc. 2020 Jun;23(6):e25544. doi: 10.1002/jia2.25544. PMID 32585077
- [Derived] Fox MP, Pascoe S, Huber AN, Murphy J, Phokojoe M, Gorgens M, Rosen S, Wilson D, Pillay Y, Fraser-Hurt N. Adherence clubs and decentralized medication delivery to support patient retention and sustained viral suppression in care: Results from a cluster-randomized evaluation of differentiated ART delivery models in South Africa. PLoS Med. 2019 Jul 23;16(7):e1002874. doi: 10.1371/journal.pmed.1002874. eCollection 2019 Jul. PMID 31335865
- [Derived] Fox MP, Pascoe SJ, Huber AN, Murphy J, Phokojoe M, Gorgens M, Rosen S, Wilson D, Pillay Y, Fraser-Hurt N. Assessing the impact of the National Department of Health's National Adherence Guidelines for Chronic Diseases in South Africa using routinely collected data: a cluster-randomised evaluation. BMJ Open. 2018 Jan 21;8(1):e019680. doi: 10.1136/bmjopen-2017-019680. PMID 29358446